CLINICAL TRIAL: NCT06690827
Title: Clinical Study of CD123 Targeting Chimeric Antigen Receptor NK Cells (CAR-NK) in the Treatment of Relapse/refractory Acute Myeloid Leukemia (AML)or Blastic Plasmacytoid Dendritic Cell Neoplasm(BPDCN)
Brief Title: Clinical Trial of CD123-targeted CAR-NK Therapy for Relapse/refractory AML or BPDCN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC065
Record Dates: First submitted 2024-11-10; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: AML (Acute Myeloid Leukemia); BPDCN (blastic Plasmacytoid Dendritic Cell Neoplasm)
Keywords: CD123; AML; Acute Myeloid Leukemia; blastic plasmacytoid dendritic cell neoplasm; acute leukemia; Malignant Hematoma; CAR-NK; CD123 CAR-NK; Chimeric antigen natural killer cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Blastic Plasmacytoid Dendritic Cell Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD123 CAR-NK cells (Experimental)
  Interventions: Drug: Anti-CD123 CAR NK cells

INTERVENTIONS:
Drug: Anti-CD123 CAR NK cells — Each patient will receive two CAR-NK cell infusions at D0 and D7, and CAR-NK cells need to be controlled within 70 minutes from thawing to infusion completion.

SUMMARY:
This is a clincal trial initiated by investigator to evaluate the safety and efficacy of anti-CD123 CAR-NK in the treatment of patients with relapsed/refractory acute myeloid leukemia or blastic plasma cell like dendritic cell tumors.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, dose-finding and expansion clinical trial aimed at evaluating the safety and efficacy of antiCD123 CAR-NK therapy for the treatment of patients with relapsed/refractory AML or BPDCN. The goal is to determine the recommended dose of CAR-NK cell therapy for these conditions. The study includes three dose groups: 1×107 CAR-positive cells/kg, 3×107 CAR-positive cells/kg, and 5×107 CAR-positive cells/kg. Each patient will receive two infusions of CAR-NK cells on D0 and D7, respectively, with the doses for both infusions principally remaining the same. However, the investigaors have the flexibility to adjust the second infusion dose based on the subject's condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any gender, aged between 18 and 75 years (inclusive);
2. Positive expression of CD123 on tumor cells detected by flow cytometry;
3. Patients with a confirmed diagnosis of CD123-positive relapsed/refractory AML or BPDCN:

(1) For AML patients：

* Relapsed refers to the reappearance of leukemic cells in peripheral blood after complete remission (CR), or ≥5% blasts in bone marrow (excluding other reasons such as bone marrow regeneration after consolidation chemotherapy), or the presence of leukemic cell infiltration outside the marrow;
* Refractory refers to patients who have not responded to two courses of standard treatment; patients who have relapsed within 12 months after CR and consolidation/intensification therapy; patients who have relapsed after 12 months but have not responded to conventional chemotherapy; patients with two or more relapses; patients with persistent extramedullary leukemia;

  (2) For BPDCN patients: Patients who have not responded to or cannot tolerate the recommended salvage treatment according to guidelines, and have persistent or recurrent disease in any of the following: peripheral blood, bone marrow, lymph nodes, spleen, skin lesions, or other sites.

  4. Expected survival time of more than 12 weeks;

  5. ECOG score of 0-2 (Appendix 2);

  6. No severe mental disorders;

  7. Basic normal function of important organs:
  1. Blood routine: white blood cells >1.0×109/L, neutrophils >0.5×109/L, lymphocytes >0.5×109/L, platelets >50×109/L;
  2. Cardiac function: echocardiography indicates a left ventricular ejection fraction ≥50%, and no significant abnormalities on electrocardiogram;
  3. Renal function: serum creatinine ≤2.0×ULN;
  4. Liver function: ALT and AST ≤3.0×ULN (for patients with liver invasion

     * 5.0×ULN);
  5. Total bilirubin ≤2.0×ULN (for patients with Gilbert's syndrome ≤3.0×ULN);
  6. Blood oxygen saturation >92%. 8. The patient or their legal guardian agrees to participate in this clinical trial and signs the ICF, indicating their understanding of the purpose and procedures of the clinical trial and willingness to participate in the study.

Exclusion Criteria:

1. Presence of active central nervous system invasion during screening;
2. Receipt of anti-tumor therapies prior to screening, including chemotherapy, targeted therapy, or other experimental drug treatments within 14 days or at least 5 half-lives (whichever is shorter), except for those who have confirmed disease progression after treatment;
3. Occurrence of cerebrovascular accident or epileptic seizure within 6 months prior to screening;
4. Presence of active or uncontrolled infection requiring systemic treatment within 1 week prior to screening;
5. Presence of any of the following cardiac diseases:

   1. Congestive heart failure at New York Heart Association (NYHA) class III or IV;
   2. Myocardial infarction or coronary artery bypass grafting (CABG) within 6 months prior to enrollment;
   3. Clinically significant ventricular arrhythmia, or history of unexplained syncope (excluding cases caused by vasovagal or dehydration);
   4. History of severe non-ischemic cardiomyopathy;
6. Combination with active autoimmune diseases requiring long-term immunosuppressive therapy;
7. Presence of other malignancies, except for adequately treated carcinoma in situ of the cervix, basal cell or squamous cell carcinoma of the skin, localized prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery.
8. Receipt of live attenuated vaccines within 4 weeks prior to screening;
9. Pregnant or breastfeeding women, as well as male or female subjects who plan to have children within 1 year after receiving CAR-NK cell infusion;
10. Other conditions that the investigator deems unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-13 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 28 dyas
  The incidence of adverse events after CAR-NK cell infusion was assessed by CTCAE, version 5.0.
Objective response rate (ORR), including complete response (CR) and partial response (PR), after CAR-NK infusion | 1month, 2 months, 3 months
overall survival (OS) after CAR-NK infusion | 2 years
Duration of response (DOR) after CAR-NK infusion | 2 years
recurrence free survival (RFS) after CAR-NK infusion | 2 years
event free survival (EFS) after CAR-NK cells infusion | 2 years

SECONDARY OUTCOMES:
Dose limited toxicity (DLT) rate after CAR-NK infusion | 1 month
Cmax of anti-CD123 CAR-NK cells in humans | 1 month
Overall response rate (ORR) after anti-CD123 CAR-NK therapy in relapsed/refractory AML and BPDCN patients | 1 year
Tmax of anti-CD123 CAR-NK cells [Cell dynamics] | 1 month
AUCs of anti-CD123 CAR-NK cells [Cell dynamics] | 1 month
overall survival (OS) after anti-CD123 CAR-NK infusion in r/r AML and BPDCN patients | 2 years
duration of response (DOR) after anti-CD123 CAR-NK cells infusion in r/r AML and BPDCN patients | 2 years
Recurrence free survival (RFS) after anti-CD123 CAR-NK cells infusion in r/r AML and BPDCN patients | 2 years
Event free survival (EFS) after anti-CD123 CAR-NK cells infusion in r/r AML and BPDCN patients | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology., Wuhan, Hubei, China